CLINICAL TRIAL: NCT06511726
Title: Induction Chemotherapy Plus Cadonilimab Followed by Chemoradiotherapy for Locally Advanced Cervical Cancer: A Multicenter, Open-label, Single-arm, Phase II Trial
Brief Title: Induction Chemotherapy Plus Cadonilimab for Locally Advanced Cervical Cancer
Acronym: CATPCC-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1101-04
Record Dates: First submitted 2024-07-11; First posted 2024-07-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; immunotherapy; Induction chemotherapy; Cadonilimab
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab plus Cisplatin and Albumin-Bound Paclitaxel as Induction therapy Followed by CCRT (Experimental): This is a single-arm study. The experimental arm includes Cadonilimab + cisplatin + albumin-bound paclitaxel, for a total of 2 cycles (cisplatin 75 mg/m² + albumin-bound paclitaxel 260 mg/m² q3w, Cadonilimab 10 mg/kg q3w).
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Induction chemotherapy and immunotherapy: Cadonilimab + cisplatin + albumin-bound paclitaxel, for a total of 2 cycles (cisplatin 75 mg/m² + albumin-bound paclitaxel 260 mg/m² q3w, Cadonilimab 10 mg/kg q3w).
  Other Names: AK-104

SUMMARY:
This is a Phase II clinical study for patients with locally advanced cervical cancer, aimed at evaluating the efficacy, safety, and tolerability of Cadonilimab combined with chemotherapy as induction therapy.

DETAILED DESCRIPTION:
This is a Phase II clinical study for patients with locally advanced cervical cancer, aimed at evaluating the efficacy, safety, and tolerability of Cadonilimab combined with chemotherapy induction therapy, as well as exploring the correlation between the expression level of PD-L1 in tumor samples, changes in blood and tumor-local immune-related factors and cells during treatment, and the efficacy of Cadonilimab induction therapy. The study is divided into two stages, with the first stage requiring the enrollment of 9 patients. If the number of effective cases is ≤7, the trial will be terminated; if >7 cases, it will proceed to the second stage, continuing to enroll patients until reaching 29. The Cadonilimab dosing regimen involves immunotherapy combined with chemotherapy induction, Cadonilimab and cisplatin and albumin-bound paclitaxel, for a total of 2 cycles. The radiotherapy and chemotherapy regimen includes cisplatin 30-40 mg/m2, once weekly for 5 times, external radiation (6MV-X-ray) at a dose of 45-60Gy/25F; and brachytherapy at a dose of 30Gy/5F. The primary endpoint of the study is ORR, with secondary endpoints being OS, PFS, and DCR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with good compliance.
2. Age ≥ 18 years (calculated on the day of signing the informed consent).
3. Histologically or pathologically diagnosed with cervical cancer (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma) and measurable lesions.
4. Initial diagnosis of stage IB3-IVA (according to FIGO 2018 staging).
5. ECOG performance score of 0-2.
6. Main organ functions meet the protocol criteria within 7 days before treatment.

Exclusion Criteria:

1. Patients with other histological types of cervical cancer, such as neuroendocrine carcinoma or sarcoma.
2. Evidence of distant metastasis, including groin lymph node metastasis and lymph node metastasis above the L1 level.
3. Previously underwent total hysterectomy (removal of the uterus body + cervix). History of subtotal hysterectomy or cervical wedge resection that preserves the cervix is allowed.
4. With anatomical abnormalities or tumor geometry-related contraindications that prevent the use of brachytherapy.
5. Within 2 years, had other active malignant tumors, except for locally curable tumors that have been cured, such as squamous cell carcinoma of the skin, basal cell carcinoma of the skin, superficial bladder cancer, and ductal carcinoma in situ of the breast.
6. With clinically significant bilateral hydronephrosis that, in the investigator's judgment, cannot be relieved by nephrostomy or ureteral stent placement.
7. Previously received immune checkpoint inhibitors (e.g., anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies) or any treatment targeting tumor immune mechanisms involving immune co-stimulatory factors (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40).
8. Within 2 weeks, requires the use of glucocorticoids (> 10 mg/day prednisone or equivalent dose of glucocorticoids) or other immunosuppressive drugs for systemic treatment exceptions include: a) Allowed treatment with inhaled, ophthalmic, or local doses ≤ 10 mg/day prednisone or equivalent dose of glucocorticoids. b) Physiological glucocorticoid replacement therapy at a dose ≤ 10 mg/day prednisone or equivalent dose of glucocorticoids. c) Glucocorticoids used for prophylaxis against hypersensitivity reactions (e.g., premedication for CT scans).
9. Within 2 weeks, received drugs with immunomodulatory effects (e.g., thymosin, interferon, interleukin-2).
10. Presence of active systemic infections requiring systemic treatment (including active pulmonary tuberculosis, active syphilis caused by Treponema pallidum, and fungal infections requiring systemic treatment) note: exclusion does not apply to antiviral drugs used for hepatitis B virus infection.
11. Within 4 weeks, experienced severe infections, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.
12. Within 4 weeks, underwent major surgical treatment (as determined by the investigator), open biopsy, or significant trauma or requires scheduled major surgical treatment during the study. Diagnostic systematic pelvic/aortic lymphadenectomy is allowed.
13. Received live vaccines within 4 weeks .
14. With active or history of documented autoimmune diseases exceptions include: vitiligo, alopecia, psoriasis, or eczema that do not require systemic treatment hypothyroidism caused by autoimmune thyroiditis requiring stable dose of hormone replacement therapy type 1 diabetes requiring stable dose of insulin replacement therapy.
15. Any of the following cardiovascular diseases: a) New York Heart Association (NYHA) functional classification ≥ II for heart failure. b) Presence of severe arrhythmias requiring long-term drug intervention asymptomatic patients with stable ventricular rate in atrial fibrillation are allowed to enroll. c) Occurrence of cerebrovascular events (CVA) within 6 months . d) Left ventricular ejection fraction (LVEF) < 50%.
16. Known primary or secondary immunodeficiency, including positive human immunodeficiency virus (HIV) antibody test.
17. Subjects with active hepatitis B virus (HBV) infection, non-active or asymptomatic carriers of hepatitis B surface antigen (HBsAg) with HBV DNA > 1000 IU/mL, and subjects with active hepatitis C virus (HCV) infection. Note: Non-active or asymptomatic carriers with treated and stable hepatitis B infection with HBV DNA ≤ 1000 IU/mL are allowed to enroll. Subjects with cured hepatitis C infection, positive HCV antibody (HCVAb), and negative HCV RNA are allowed to enroll.
18. With active or documented history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis) or active diverticulitis.
19. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
20. Known history of severe hypersensitivity reactions to other monoclonal antibodies.
21. Pregnant or breastfeeding women.
22. The investigator believes that there may be risks associated With receiving the investigational drug or any condition that may interfere With the evaluation of the investigational drug, subject safety, or interpretation of study results (such as having other severe diseases or mental disorders).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to18 months
  At 2 weeks post-induction therapy, objective response rate represents the proportion of patients showing a predefined level of tumor shrinkage or disappearance in response to treatment.

SECONDARY OUTCOMES:
OS | up to approximately 46 months
  Overall survival measures the length of time from the start of treatment until death from any cause, indicating the effectiveness of the treatment in prolonging patients' lives.
PFS | up to approximately 46 months
  Progression-free survival measures the length of time during and after treatment that a patient lives with the disease without it progressing.
DCR | up to approximately 46 months
  DCR is the proportion of patients who have achieved complete response, partial response, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Shoumin Bai, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial hosipital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No